CLINICAL TRIAL: NCT02675413
Title: Mechanisms of Action of Dimethyl Fumarate in Relapsing MS
Brief Title: Mechanisms of Action of Dimethyl Fumarate (Tecfidera) in Relapsing MS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator decided to withdraw.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201511112
Record Dates: First submitted 2016-01-11; First posted 2016-02-05 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Cerebral Spinal Fluid; Dimethyl Fumarate; Tecfidera; Multiple Sclerosis; Relapsing MS; RRMS; Mechanism of Action
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dimethyl Fumarate (Experimental): Open label dimethyl fumarate (Tecfidera) at the US approved dose of 120mg BID for 7 days and then 240mg BID thereafter for 12 months.
  Interventions: Drug: Dimethyl Fumarate

INTERVENTIONS:
Drug: Dimethyl Fumarate — Open-label
  Other Names: Tecfidera

SUMMARY:
This is a prospective study that will explore the mechanisms of efficacy of dimethyl fumarate (DMF) treatment in multiple sclerosis (MS). Investigators will enroll relapsing MS patients who are beginning therapy with DMF into a one-year longitudinal study in which blood and spinal fluid analyses, imaging and clinical studies will be performed to identify and measure changes associated with DMF therapy.

DETAILED DESCRIPTION:
The emergence of Dimethyl Fumarate (DMF) as an oral agent for the treatment of relapsing multiple sclerosis (MS) has the potential to reduce the burden of neurologic disability while minimizing side effects and risks associated with more established therapies. However, at present there is a need for further understanding of the mechanisms of action for DMF. That is, it is not yet known whether the benefits observed in MS patients treated with DMF are due primarily to immunologic and anti-inflammatory effects or neuroprotective effects, or both. The main site(s) of DMF actions, whether in the CNS and/or the periphery, is also not known.

Dimethyl fumarate is believed to act centrally by enhancing the nuclear factor erythroid 2 related factor 2 (Nrf2) transcriptional pathway, which regulates enzymes to counter act oxidative stress . DMF may enhance the Nrf2 transcriptional pathway within the CNS, but this is unproven. DMF is also anti-inflammatory, and is known to inhibit NFB translocation to the nucleus [and chemokine-induced monocyte chemotaxis. Inhibition of NFB could occur systemically, or within the CNS, or both. Therefore, investigators intend to investigate antioxidant and immunologic changes within the central nervous system (CNS) and blood in relation to DMF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsing MS (2010 McDonald Criteria)
* Age greater than or equal to 18.
* Starting treatment with dimethyl fumarate (DMF). Enrolled patients will be either naive to disease modifying therapy (DMT) or will be enrolled after a greater than or equal to 30 days from last dose of prior DMT. If enrolled patients cannot tolerate DMF, the will be replaced by another subject. All subjects will serve as their own control.

Exclusion Criteria:

* Women of Childbearing Potential who are pregnant, breastfeeding, or planning to become pregnant or breastfeed for the duration of the study.
* Chronic diseases that will have effects on the laboratory, clinical and imaging parameters we will study: Insulin-dependent diabetes mellitus, stroke, Alzheimer's disease, auto-immune disorders such as rheumatoid arthritis, lupus, neuromyelitis optica, mixed connective disease, or sjogren's disease.
* Any prior treatment with mitoxantrone or alemtuzumab.
* Those undergoing DMT within the past 12 months with rituximab or daclizumab.
* Patients treated with chronic (monthly) systemic steroids.
* Patients treated with steroids (intravenous, intramuscular, oral or ACTH) with the intent to treat MS within 30 days of the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean differences in Indicators of Oxidative stress (Nitrate, nitrite (um/L), Glutathione (uM), and F2-isoprostanes (pg/ml)) in blood and CSF at baseline and 12 months | 24 months
  Mean difference in Nitrate, nitrite (um/L), Glutathione (uM), and F2-isoprostanes (pg/ml)
Mean differences in markers of axonal damage to assess whether DMF protects against neurodegeneration at baseline and 12 months | 24 months
  mean differences in neurofilament heavy and light chains, and tau protein in blood and spinal fluid
Mean differences in MS-relevant cytokines, chemokines and osteopontin to examine the immunologic consequences of DMF therapy during autoimmune CNS inflammation. | 24 months
  Mean differences in CXCL13 (pg/ml), CCL2 (pg/ml), TNF (pg/ml), IFNg (pg/ml),IL-17 (pg/ml), Osteopontin (pg/ml)
Mean differences in the phenotype and activation status of adaptive and innate immune cells in the CSF and peripheral circulation at baseline and 12 months. | 24 months
  Mean differences in CD4 (% and cells/uL) , CD8 (% and cells/uL), CD117 (% and cells/uL), HLA-DR (% and cells/uL), CD123 (% and cells/uL), CD19 (% and cells/uL),CD14, monocytes (% and cells/uL), CD11c (% and cells/uL), BDCA2 (% and cells/uL), CD56 and CD16, NK cells (% and cells/uL), CD138, plasmablasts (% and cells/uL)

SECONDARY OUTCOMES:
Correlation of Biomarkers with Imaging and Clinical Outcome Measures | 24 months
  A secondary goal is to correlate the biomarkers listed in the primary objectives with the number of gadolinium enhancing, T2W and T1W lesions seen at baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cross, MD, Principal Investigator — Washington University School of Medicine; Laura Piccio, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University (John L. Trotter MS Center), St Louis, Missouri
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Unclear what results may be available for sharing. We plan to publish group analysis.